CLINICAL TRIAL: NCT02910453
Title: VATS Versus Open Pulmonary Lobectomy for Lung Cancer: a Prospective Analysis of Different Impacts on Ribcage Kinematics With Optoelectronic Plethysmography
Brief Title: VATS Versus Open Pulmonary Lobectomy in the Limelight of OEP
Acronym: VOLO
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Sponsor
Other Study IDs: VOLO-2016-2583
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2016-09

CONDITIONS: Lung Cancer
Keywords: Pulmonary lobectomy; Video-Assisted Thoracic Surgery; Opto-electronic plethysmography; Posterolateral thoracotomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- VATS group: Pulmonary lobectomy via VATS. VATS starts with a utility incision, approximately 4 cm in length, anterior to the latissimus dorsi muscle at the 4th intercostal space. Muscle fibers are split without cutting and a wound protector is regularly placed in site. The camera port is placed in the 6th or 7th intercostal space at the anterior axillary line and a third 10-mm access is made at the same intercostal space at the posterior axillary line. The hilum is approached anteriorly
  Interventions: Procedure: Pulmonary lobectomy
- Open group: Pulmonary lobectomy via posterolateral thoracotomy (PLT). PLT consists in a standard 10-15 muscle-sparing incision at 4th intercostal space, rib divaricators are utilized and the hilum is approached posteriorly as previously described
  Interventions: Procedure: Pulmonary lobectomy

INTERVENTIONS:
Procedure: Pulmonary lobectomy

SUMMARY:
The standard operative approach to pulmonary lesions has been via postero-lateral thoracotomy and direct vision. This technique has some advantages but its morbidity is significant. Some surgeons advocate a resection by video-assisted thoracic surgery (VATS) to reduce the impact on chest wall and the impairment on respiratory mechanic. However, an evidence for superiority of the approach minimally invasive is lacking, particularly for the difficult assessment of the change in pulmonary function. The aim of this study is to compare VATS- over open lobectomy regarding the differences of chest wall kinematic, analyzed by optoelectronic plethysmography (OEP).

DETAILED DESCRIPTION:
Rationale: The standard operative approach to pulmonary lesions has been via postero-lateral thoracotomy and direct vision. This technique has some advantages but its morbidity is significant. Some surgeons advocate a resection by video-assisted thoracic surgery (VATS) to reduce the impact on chest wall and the impairment on respiratory mechanic. However, an evidence for superiority of the approach minimally invasive is lacking, particularly for the difficult assessment of the change in pulmonary function and its relation with chest wall modifications.

Objective: The aim of this study is to compare VATS- over open lobectomy regarding the differences of chest wall kinematic analyzed by optoelectronic plethysmography (OEP).

Study design: A prospective mono-centre single blind trial. Study population: Adult patients of either gender candidate for pulmonary lobectomy for non small cell lung cancer.

Intervention: Patients are submitted to pulmonary lobectomy by video-assisted technique or by postero-lateral thoracotomy. This decision follows the usual clinical evaluations, regardless of whether or not the study enrollment. In particular, they are candidates for postero-lateral thoracotomy if: tumors were close to the hilum or other relevant anatomical structures, or the computed tomography demonstrated hilar calcific lymph-nodes or the lesions were of greater than 4 cm diameter.

Endpoint is evaluation of modification of respiratory kinematic after pulmonary lobectomy, assessed by OEP. In particular, the volume variation of pulmonary rib cage of the treated side versus the relative untreated side and the differences. Respiratory movements and thoracic and abdominal volume changes will be recorded continuously by analyzing the movements of retro-reflective markers using 8 video-cameras connected to an automatic optoelectronic motion analyzer. Subjects are prepared for OEP (markers). Baseline spirometry is take prior to exercise test. All exercise take place on an electromagnetically braked cycle-ergometer. Throughout the protocol heart rate, oxygen saturation and dyspnoea with the Borg scale are recorded. Ventilatory kinematics are monitored throughout exercise using OEP. This OEP analysis involves compartmentalization of the chest into three sections: pulmonary rib cage, abdominal rib cage, and abdomen to determine the contribution of each component to total chest wall volume.

ELIGIBILITY:
Inclusion Criteria:

* Lesion not in close relation to the hilar structures (bronchus, vessels) based on CT
* Non-Small Cell Lung Cancer clinically staged T1-2, N0 or N1, M0
* Subject must be able to tolerate general anesthesia and have cardiopulmonary reserve to tolerate a lobectomy

Exclusion Criteria:

* Previous thoracic surgery on same side
* Planned segment resection or pneumonectomy
* Any type of chronic pain, requiring daily use of analgesics
* Body Mass Index (BMI) ≥ 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients suitable for pulmonary lobectomy.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Modification of respiratory kinematic | T0: preoperatively (2 weeks before surgery); T1: 1 week after surgery; T2: 2 months after surgery
  Compare VATS- over open pulmonary lobectomy regarding the differences of chest wall kinematic, analyzed by optoelectronic plethysmography (OEP)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Derived] LoMauro A, Aliverti A, Chiesa M, Cattaneo M, Privitera E, Tosi D, Nosotti M, Santambrogio L, Palleschi A. Ribcage kinematics during exercise justifies thoracoscopic versus postero-lateral thoracotomy lobectomy prompt recovery. Eur J Cardiothorac Surg. 2017 Dec 1;52(6):1197-1205. doi: 10.1093/ejcts/ezx174. PMID 28977548